CLINICAL TRIAL: NCT02304354
Title: Relationship Between T LYmphocytes Depletion and Clinical Response to RITUXimab in Rheumatoid Arthritis (LYRITUX)
Acronym: LYRITUX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRI13-JM/LYRITUX; 2014-000859-91 (EudraCT Number); 2014-R24 (Other: CPP); 140896A-32 (Other: ANSM)
Record Dates: First submitted 2014-11-04; First posted 2014-12-01 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; T lymphocytes; rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): two intravenous infusions of 1000 mg with a two-week interval between them
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — For rheumatoid arthritis, MabThera is given as two intravenous infusions of 1000 mg with a two-week interval between them. Patients usually respond to treatment within 16 to 24 weeks of initial treatment. After 24 weeks, treatment can be repeated depending on the patient's response.
  Other Names: MabThera

SUMMARY:
Rituximab, an anti CD-20 monoclonal antibody targeting B lymphocytes is prescribed in rheumatoid arthritis (RA) patients refractory to TNF alpha antagonists. According to previous studies, 25 to 50% of patients have an insufficient or absence of response to rituximab at week 24.

In a recent retrospective study, a CD4+ T-lymphocytes depletion was observed after a first course of rituximab in RA patients. The absolute CD4+ number at week 12 was 37% (±33) of the baseline value, leading to < 200 cells/µL in 5% of patients. Interestingly the absence of CD4+ T-lymphocytes depletion was observed in clinical non-responders, suggesting the involvement of T-lymphocytes in the mechanism of action of rituximab. So far no prospective study have supported the usefulness of lymphocyte phenotyping, in particular T-lymphocytes, to monitor rituximab-treated RA patients.

DETAILED DESCRIPTION:
Rituximab, an anti CD-20 monoclonal antibody targeting B lymphocytes is prescribed in rheumatoid arthritis (RA) patients refractory to TNF alpha antagonists. According to previous studies, (Edwards, Szczepanski et al. 2004; Cohen, Emery et al. 2006; Emery, Fleischmann et al. 2006) 25 to 50% of patients have an insufficient or absence of response to rituximab at week 24. In the pathogenesis of RA, B and T lymphocytes are tightly linked through the APC fonction and cytokines production of B lymphocytes. At present, a white blood cells count is recommended in routine every 3 months in patients receiving rituximab, since cases of neutropenia have been observed in approximately 8% of patients with lymphoma after treatment. In RA patients, B lymphocytes count before each rituximab course should be done to prevent opportunistic infections (Pham, Fautrel et al. 2008).

In a recent retrospective study, a CD4+ T-lymphocytes depletion was observed after a first course of rituximab in RA patients. The absolute CD4+ number at week 12 was 37% (±33) of the baseline value, leading to < 200 cells/µL in 5% of patients. Interestingly the absence of CD4+ T-lymphocytes depletion was observed in clinical non-responders, suggesting the involvement of T-lymphocytes in the mechanism of action of rituximab (Mélet, Mulleman et al. 2013). Moreover, few case reports of RA patients developing opportunist infections in conjunction with CD4+ T-lymphocyte depletion have been published (Teichmann, Woenckhaus et al. 2008; Clifford, Ances et al. 2011). So far no prospective study have supported the usefulness of lymphocyte phenotyping, in particular T-lymphocytes, to monitor rituximab-treated RA patients.

ELIGIBILITY:
Inclusion Criteria:

* RA according to the American College of Rheumatology (ACR) criteria
* Treatment with adalimumab in accordance to the SPC
* Disease modifying anti rheumatic drugs (DMARDs) stable 4 weeks before enrollment and during 16 weeks.
* Signed consent

Exclusion Criteria:

* No anti TNF-alpha failure or contraindication
* Previous adalimumab treatment
* Contraindication to adalimumab, methylprednisolone or methotrexate (when used in combination with adalimumab)
* methotrexate-naive patient
* Any hematologic disease affecting the lymphocytes (in particular lymphomas)
* Any osteo-articular disease which could interfere with the interpretation of the influence of the rituximab on RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
DAS28 | up week 48
  Disease Activity Score on 28 joints (DAS28) is a composite score that comprise tender joints count, swollen joints count, patient's disease activity on visual analog scale and erythrocyte sedimentation rate. DAS28 will be measured at baseline, week 2, week 4, week 16 and at the end of the study (i.e. between week 24 and week 48).
T-lymphocyte count | up to week 48
  T-lymphocyte count will be measured at baseline, week 2, week 4, week 16 and at the end of the study (i.e. between week 24 and week 48).

SECONDARY OUTCOMES:
C reactive Protein (CRP) | Baseline up to 48 weeks
  CRP will be measured at baseline, week 2, week 4, week 16 and at the end of the study (i.e. between week 24 and week 48).
Immunoglobulines G | Baseline up to 48 weeks
  Immunoglobuline G concentrations will be measured at baseline, week 16 and at the end of the study (i.e. between week 24 and week 48).
Cytokine profile | Baseline up to 48 weeks
  the following cytokines (APRIL, BAFF, TNF, IL-1 alpha, IL-17 and IL-6) will be measured at baseline, week 2, week 4, week 16 and at the end of the study (i.e. between week 24 and week 48).
Occurrence of infections | Baseline up to 48 weeks
  Number of participants with infectious adverse events
Pharmacokinetics (Systemic Clearance and central volume of distribution) | Baseline up to 48 weeks
  Rituximab concentrations will be measured at baseline, will be measured at baseline, week 2, week 4, week 16 and at the end of the study (i.e. between week 24 and week 48). Pharmacokinetics will be described using a two-compartment model.
FCGR3A 156 F/V gene polymorphism | Baseline
  FCGR3A 156 F/V gene genotyping. Measurements will be carried out at baseline.
RNA | Baseline
  Gene expression will be analysed at baseline.
Metabolomic profil | Baseline up to 16 weeks
  Urines will be analysed at baseline, week 4 and week 16

CONTACTS AND LOCATIONS:
Overall Officials: Denis MULLEMAN, MD-PhD, Principal Investigator — CHRU de TOURS
Locations (8):
- France (8):
  - Rhumatologie, CHRU de BREST, Brest
  - Rhumatologie, CHD LA ROCHE SUR YON, La Roche-sur-Yon
  - Rhumatologie, CHR du MANS, Le Mans
  - Rhumatologie, CHRU de NANTES, Nantes
  - Rhumatologie / IPROS, CHR d'ORLEANS, Orléans
  - Rhumatologie, CHRU de POITIERS, Poitiers
  - Rhumatologie, CHRU de ROUEN, Rouen
  - Rhumatologie, CHRU de TOURS, Tours

REFERENCES:
- [Background] Melet J, Mulleman D, Goupille P, Ribourtout B, Watier H, Thibault G. Rituximab-induced T cell depletion in patients with rheumatoid arthritis: association with clinical response. Arthritis Rheum. 2013 Nov;65(11):2783-90. doi: 10.1002/art.38107. PMID 23918413